CLINICAL TRIAL: NCT05282511
Title: Identification of the Key Factors Increasing the Risk of Vasospastic Angina Based on Multi-omics.
Brief Title: A Multi-Omics Study of Vasospastic Angina
Acronym: KIVAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Dao Wen Wang, Prof, Tongji Hospital
Other Study IDs: JTH-KIVAM
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Vasospastic Angina
MeSH Terms: conditions — Angina Pectoris, Variant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Serum, Blood Cells and DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with acute myocardial infarction: Patients with acute myocardial infarction
- Healthy controls: Healthy controls
- Patients with vasospastic angina: Patients with vasospastic angina

SUMMARY:
This is a observational study to identify the key factor associated with vasospastic angina and to explore the prognosis of the participants. The study will recruit 400 patients with vasospastic angina, 400 healthy controls and 400 patients with acute myocardial infarction. Next generation sequencing, metabolome and proteomics will be performed in these participants.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* diagnosed as vasospastic angina

Exclusion Criteria:

* participate in any drug clinical trials within 3 months
* patients with life-threatening complications, or the researchers determined that the survival time of patients with no more than 1 years
* serious neurological disease (Alzheimer's disease, Parkinson syndrome, progressive lower limbs or deaf patients)
* previous history of cancer or tumor, or pathological examination confirmed precancerous lesions (such as breast ductal carcinoma in situ, or atypical hyperplasia of the cervix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chinese patients with vasospastic angina
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2012-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Death | up to 48 months
  Death from cardiovascular causes and any unknown death unless there was another certain cause
Stroke | up to 48 months
  A rapid onset of a new focal loss of neurologic function caused by an ischemic central nervous system event with residual symptoms lasting at least 24 hours from their onset or leading to death
Myocardial Infarction | up to 48 months
  The definition of myocardial infarction was consistent with the Third Universal Definition of Myocardial Infarction.

SECONDARY OUTCOMES:
Recurrent angina | up to 48 months
  Recurrent angina
Rehospitalization due to cardiovascular causes | up to 48 months
  Rehospitalization due to cardiovascular causes

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China